CLINICAL TRIAL: NCT00446719
Title: An Open-Label Pilot Study Evaluating the Safety and Antidepressant Effects of Rellidep (BI= Biological Isolate) in Major Depressive Disorder
Brief Title: Safety and Antidepressant Effects of Rellidep in Major Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Joel Sadavoy MD. Head community psychiatry and geriatric psychiatry programs, 600 university Ave Toronto M5G 1X5
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSH 06-0307-A
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Depression
Keywords: major depression; antidepressant; quality of life; anxiety
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Anxiety Disorders | interventions — rellidep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rellidep — 2000 mg P.O. daily for 8 weeks

SUMMARY:
The investigators hypothesize that Rellidep will be effective in improving the symptoms of major depression. The available evidence strongly suggests that Rellidep contains a mood altering ingredient or ingredients. This open-label, non-randomized study sets out to validate its potential antidepressant activity.The study will include secondary aims of evaluating the effect of Rellidep on reducing symptoms of anxiety, a common symptom associated symptom of depression and improving quality of life.

About twenty-five patients with major depressive disorder will be assigned to open-label Rellidep (2000 mg/day) for a period of 8 weeks. All patients will be assessed by various measures of global improvement, depression, quality of life, sexual experience, anxiety and measures of side effects as well as standard laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained.
* Males/Females 20-65 years of age who require a new or a new change in their medication treatment for diagnosed major depression.
* A clinical diagnosis fulfilling DSM-IVTR criteria for Major Depressive Disorder, single episode or recurrent.
* 17-Item Hamilton Depression Rating Scale (HAMD 17-item) total score at baseline of 18 or higher

Exclusion Criteria:

* Clinical diagnosis of depression other than DSM-IVTR Major Depressive Disorder (single episode/recurrent, e.g. chronic depression and/or refractory depression are excluded).
* Judged to be at significant risk for suicide or having a history suggesting significant current potential for self harm.
* Antidepressant medication (other than the index antidepressant).
* Women who are pregnant or breast-feeding or intending to become pregnant in the next 12 months.
* Clinically significant organ system diseases, e.g. cardiovascular, hepatic, renal, endocrine, gastrointestinal, metabolic, or other systemic diseases.
* Course of electroconvulsive therapy (ECT) during the observational period.
* Suffer from a major neurological condition (i.e., Parkinson's disease, Huntington's disease), cerebrovascular disease (i.e., stroke), metabolic conditions (i.e., Vitamin B12 deficiency), autoimmune conditions (i.e., systematic lupus erythematosus), viral or other infections (i.e., hepatitis, mononucleosis, human immunodeficiency), and cancer.
* Current diagnosis of Schizophrenia or other psychotic disorders (including Schizophreniform Disorder, Schizoaffective Disorder, Delusional Disorder, brief psychotic disorders, psychotic disorder due to general medical condition, substance induced psychotic, psychotic disorder not otherwise specified) as defined in the DSM-IV.
* (Sub) clinical hypo/hyper thyroidism (e.g. elevated TSH).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
50% improvement on Hamilton Depression Rating Scale-17 at 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Clinical Global Impression-Severity and Improvement | 8 weeks
Montgomery Asberg Depression Rating Scale (MADRS) at 8 weeks | 8 weeks
Medical Outcomes Study Short-Form 36 (SF-36)at 8 weeks | 8 weeks
Beck Depression Inventory Scale (BDI) a t 8 weeks | 8 weeks
Hamilton rating scale for Anxiety (HAM-A)at 8 weeks | 8 weeks
UKU | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel Sadavoy M.D., Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada